CLINICAL TRIAL: NCT05123339
Title: Clinical Signs and Activity Limitations Associated With Dural Ectasia in Patients With Marfan Disease: Cross-sectional Case-control Study.
Brief Title: Clinical Signs and Activity Limitations Associated With Dural Ectasia in Patients With Marfan Disease
Acronym: MARFANLOMB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211106; 2021-A00654-37 (Other: France : Ministry of Health)
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Marfan Syndrome
Keywords: Marfan's disease; Dural ectasia; Clinical signs; Intracranial hypotension; Low back pain; Activity limitation
MeSH Terms: conditions — Marfan Syndrome; Arachnodactyly; Signs and Symptoms; Intracranial Hypotension; Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Marfan disease according to Ghent criteria revised in 2010 with dural ectasia Patients followed at the CNMR in Bichat Adults ≥18 years old and ≤ 55 years old (to limit the incidence of degenerative lumbar pathologies) No history of lumbar surgery <1 year and without specific pathologies of the spine (tumor, infection, trauma, fracture, inflammatory rheumatism)
  Interventions: Other: Questionnaire
- Control group: Marfan disease according to Ghent criteria revised in 2010 without dural ectasia Patients followed at the CNMR in Bichat Adults ≥18 years old and ≤ 55 years old (to limit the incidence of degenerative lumbar pathologies) No history of lumbar surgery <1 year and without specific pathologies of the spine (tumor, infection, trauma, fracture, inflammatory rheumatism)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
Primary outcome is to compare the frequency and clinical features of spinal symptoms between Marfan patients with dural ectasia (cases) and those without (controls).

1. / Frequency of orthostatic headaches
2. / Frequency of low back pain due to orthostasis
3. / Frequency of low back pain during Vasalva maneuvers
4. / Frequency of lumbar claudication
5. / Frequency of root claudication

Secondary outcomes are to compare activity limitations, quality of life and intensity of low back and radicular pain between Marfan patients with dural sac ectasia (cases) and those without (controls).

1. / Average intensity of back pain measured on a self-administered digital scale (0 = no pain and 100 = maximum pain)
2. / Average intensity of radicular pain measured on a self-administered digital scale (0 = no pain and 100 = maximum pain)
3. / Activity limitations specific to the lumbar spine measured using the self-administered Oswestry Disability Index questionnaire (ODI, 0 = no limitations and 100 = maximum limitations)
4. / Physical component of quality of life measured using the physical component of the self-administered questionnaire 12-Item Short Form Health Survey (SF-12, 9.95 = worst quality of life imaginable, 70.02 = worst quality of life imaginable )
5. / Mental component of the quality of life measured using the mental component of the SF-12 self-administered questionnaire (5.89 = worst quality of life imaginable, 71.97 = worst quality of life imaginable)

DETAILED DESCRIPTION:
Marfan's disease is a rare condition. Clinical phenotypes are heterogeneous. Among the abnormalities of the spine, dural ectasia is common with a prevalence of 66%. This is a major sign of Ghent's diagnostic criteria. To our knowledge, the clinical and functional signs associated with dural sac ectasia have never been described with precision. Only a few uncontrolled case series have been published. This is the case of the study by Foran and colleagues published in the American Journal of Genetics in 2005 which included 22 patients with Marfan disease with dural ectasia questioned about their symptoms and quality of life. We hypothesize the existence of a clinical and functional spinal phenotype specific to dural ectasia in patients with Marfan disease.

ELIGIBILITY:
Inclusion Criteria:

* Marfan disease according to the Ghent criteria revised in 2010
* Patients followed at the CNMR in Bichat
* Adults ≥18 years old and ≤ 55 years old (to limit the incidence of degenerative lumbar pathologies)
* Patient not opposing the research
* Mastery of the French language

Exclusion Criteria:

* History of lumbar surgery <1 year
* Specific pathologies of the spine (tumor, infection, trauma, fracture, inflammatory rheumatism)
* Inability to write, read or speak French
* Cognitive or behavioral problems making assessment impossible
* Patients receiving AME
* Patients under tutorship or curatorship

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients screened and selected at the CNMR at Bichat Hospital will receive a letter containing the information note and a self-questionnaire to complete.
  Patients can reach Dr Troussier by phone or email to ask any questions. Patients will return a copy of the completed briefing note and self-questionnaire by post.
  In the event of the presence of dural sac ectasia, patients will also be asked to send in the reply letter a copy of an imaging report, MRI or lumbar CT or TAP, or failing that an account- medical report mentioning this presence.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Frequency of spinal symptoms | Inclusion
  Frequency of spinal symptoms between Marfan patients with dural ectasia (cases) and those without (controls) :
  1. / Frequency of orthostatic headaches
  2. / Frequency of low back pain due to orthostasis
  3. / Frequency of low back pain during Vasalva maneuvers
  4. / Frequency of lumbar claudication
  5. / Frequency of root claudication

SECONDARY OUTCOMES:
Self-administered digital scale (0 = no pain and 100 = maximum pain) | Inclusion
  Intensity of low back pain between Marfan patients with dural ectasia (cases) and those without (controls) : average intensity of back pain measured on a self-administered digital scale (0 = no pain and 100 = maximum pain)
Self-administered digital scale (0 = no pain and 100 = maximum pain) | Inclusion
  Intensity of radicular pain between Marfan patients with dural ectasia (cases) and those without (controls) : average intensity of radicular pain measured on a self-administered digital scale (0 = no pain and 100 = maximum pain)
Oswestry Disability Index questionnaire (ODI, 0 = no limitations and 100 = maximum limitations) | Inclusion
  Limitations between Marfan patients with dural ectasia (cases) and those without (controls) : activity limitations specific to the lumbar spine measured using the self-administered Oswestry Disability Index questionnaire (ODI, 0 = no limitations and 100 = maximum limitations)
12-Item Short Form Health Survey (SF-12, 9.95 = worst quality of life imaginable, 70.02 = worst quality of life imaginable ) | Inclusion
  Quality of life between Marfan patients with dural ectasia (cases) and those without (controls) : physical component of quality of life measured using the physical component of the self-administered questionnaire 12-Item Short Form Health Survey (SF-12, 9.95 = worst quality of life imaginable, 70.02 = worst quality of life imaginable )
12-Item Short Form Health Survey (SF-12, 9.95 = worst quality of life imaginable, 70.02 = worst quality of life imaginable ) | Inclusion
  Quality of life between Marfan patients with dural ectasia (cases) and those without (controls) : mental component of the quality of life measured using the mental component of the SF-12 self-administered questionnaire (5.89 = worst quality of life imaginable, 71.97 = worst quality of life imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle NGUYEN, Dr, Principal Investigator — Rehabilitation Service of the Musculoskeletal System and Spine Pathologies - Cochin Hospital - Paris
Locations (1):
- CNMR Bichat, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boker T, Vanem TT, Pripp AH, Rand-Hendriksen S, Paus B, Smith HJ, Lundby R. Dural ectasia in Marfan syndrome and other hereditary connective tissue disorders: a 10-year follow-up study. Spine J. 2019 Aug;19(8):1412-1421. doi: 10.1016/j.spinee.2019.04.010. Epub 2019 Apr 15. PMID 30998996
- [Background] Chuzel Q, Dupuis-Girod S, Rousset M, Decharry C, Decullier E, Pialat JB. Assessment of Dural Ectasia Using Computed Tomodensitometry as a Criterion in Marfan Syndrome. J Comput Assist Tomogr. 2019 Mar/Apr;43(2):282-287. doi: 10.1097/RCT.0000000000000822. PMID 30371622
- [Background] Foran JR, Pyeritz RE, Dietz HC, Sponseller PD. Characterization of the symptoms associated with dural ectasia in the Marfan patient. Am J Med Genet A. 2005 Apr 1;134A(1):58-65. doi: 10.1002/ajmg.a.30525. PMID 15690402
- [Background] Nguyen C, Papelard A, Schnitzler A, Mangione P, Poiraudeau S, Rannou F. Congenital lumbar spinal stenosis associated with Marfan syndrome. Joint Bone Spine. 2012 Mar;79(2):199-200. doi: 10.1016/j.jbspin.2011.07.007. Epub 2011 Oct 1. No abstract available. PMID 21962385
- [Background] Troussier S, Milleron O, Rannou F, Eliahou L, Jondeau G, Nguyen C. Painful symptoms and spine-specific activity limitations associated with dural ectasia in individuals with Marfan syndrome: a cross-sectional comparative study (MARFANLOMB). Eur Spine J. 2025 Aug;34(8):3087-3094. doi: 10.1007/s00586-025-08911-z. Epub 2025 May 31. PMID 40450135